CLINICAL TRIAL: NCT01569191
Title: Investigating the Efficacy of Artificial Tear Supplements and Cold Compresses for the Treatment of Seasonal Allergic Conjunctivitis
Brief Title: Non-Pharmaceutical Treatment of Seasonal Allergic Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aston University (Other)
Collaborators: University of Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Allergy12
Record Dates: First submitted 2012-03-27; First posted 2012-04-03 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2015-07

CONDITIONS: Hypersensitivity
Keywords: Ocular allergy; Tear supplement; Cold compress
MeSH Terms: conditions — Hypersensitivity | interventions — epinastine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- No Treatment (No Intervention): Exposure to grass pollen only
- Artificial Tear Supplement (Active Comparator): Preservative free Hypromellose Eye Drops BP 0.3% w/v preservative free - MHRA product licence number:23097/0006
  Interventions: Other: Artificial Tear Supplement
- Cold compress (Active Comparator): Cooled gel eye mask http://www.visiondirect.co.uk/vision-direct/eye-gel-mask-blue
  Interventions: Device: Cold compress
- Anti-allergic Medication (Active Comparator): ELESTAT® (epinastine HCl ophthalmic solution) 0.05% Initial U.S. Approval: 2003 H1 histamine receptor antagonist indicated for the prevention of itching associated with allergic conjunctivitis
  Interventions: Drug: Anti-allergic Medication

INTERVENTIONS:
Other: Artificial Tear Supplement — artificial tear supplement (Hypromellose)
  Other Names: Hypromellose is also sold as Isopto plain eye drops
  Arms: Artificial Tear Supplement
Device: Cold compress — Cold compress bag fill with temperature retention gel placed over closed eyes Sold by http://www.visiondirect.co.uk/vision-direct/eye-gel-mask-blue
  Other Names: Eye-gel-mask-blue
  Arms: Cold compress
Drug: Anti-allergic Medication — 1 drop on single occasion after exposure to grass pollen
  Other Names: ELESTAT® (epinastine HCl ophthalmic solution) 0.05%
  Arms: Anti-allergic Medication

SUMMARY:
Seasonal allergic conjunctivitis (SAC) is an irritating eye condition that affects many people, caused by hypersensitivity to normally harmless substances such as pollen, and often accompanies seasonal hay fever. Treatments that can be used before initiating medical therapy include artificial tear supplements (ATS) and cold compresses (CC). However, there is no evidence in the scientific literature that demonstrates their efficacy compared to no treatment or their combined effect with anti-allergic medication. Therefore the investigators aim to examine the efficacy of ATS and CC alone, in comparison to anti-allergic medication, and CC in combination with anti-allergic medication. In addition, the investigators also aim to determine the time course of ocular allergic reactions. At the end of the study the investigators will be able to see whether or not ATS and CC are effective in treating SAC.

DETAILED DESCRIPTION:
There will be a total of 6 study visits, each lasting approximately 1 hour and separated by at least 2 days. At the beginning of each visit, a set of measurements will be taken by an experienced optometrist. These are:

* What symptoms you are feeling and how severe they are - you will be asked to complete a short questionnaire about how your eyes currently feel.
* The redness and temperature of your eyes - the front surface of both eyes will be photographed using digital cameras.

After these measurements we will ask you to stand inside a specially designed room where the environment can be controlled by a computer. The pollen that you were found to be allergic to will then be introduced into the atmosphere of the room, so that the signs and symptoms of SAC can be induced - this is intentional, but normally resolves within a few hours with no treatment. At each visit, you will experience a different duration (no longer than 10 minutes) and either no treatment, artificial tear supplement (ATS; preservative free ocular lubricant), cold compress (CC; cooled gel eye mask) or anti-allergic medication (epinastine hydrochloride 500μg/mL). The measurements will then be repeated even 5 minutes for an hour.

After the final set of measurements, the front surface of your eyes will be assessed using a temporary dye to highlight using a blue light any changes. Fluorescein dye does not sting, lasts only a few minutes and has no effect on vision or driving. However it may cause a self limiting mild allergic reaction where the eyes become red, irritated and sore but this is highly unlikely as there are no known reported cases. In the unlikely event this does happen the experienced optometrist is immediately available to manage the condition.

The anti-allergic drug epinastine hydrochloride (Elestat, Allergan) is a prescription only medicine indicated for the treatment of allergic conjunctivitis. As with all medications, there are potential side effects - although uncommon (1 in 10 to 1 in 100 people), there may be a slight burning sensation on application but this temporary and subsides quickly. The epinastine formulation also contains preservatives called benzalkonium chloride and disodium edetate. As with fluorescein sodium, these may cause a self limiting mild allergic reaction. In the unlikely event this does happen the experienced optometrist is immediately available to manage the condition.

Study Length and Reimbursement Each of the 6 measurement visits is separated by 7 days therefore the total study length for each participant is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* history of seasonal allergic conjunctivitis or seasonal allergic rhinoconjunctivitis (seasonal hay fever) that is not currently active.

Exclusion Criteria:

* eye surgery in the last 3 months
* active eye condition
* adverse reaction to ocular drugs or dyes
* history of anaphylaxis (severe systemic allergic reaction)
* use any ocular medication or systemic medications (antihistamines, mast cell stabilisers, non-steroidal anti-inflammatory drugs or steroids) at least 14 days prior to the start and for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Wolffsohn, PhD, Principal Investigator — Aston University
Locations (1):
- National Pollen and Aerobiology Unit, Worcester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- No Treatment/Artificial Tear / Cold Compress / Pharmaceutical: Exposure to grass pollen only
  Preservative free Hypromellose Eye Drops BP 0.3% w/v preservative free - MHRA product licence number:23097/0006 Non-Pharmaceutical Tear Supplement artificial tear
  Cooled gel eye mask http://www.visiondirect.co.uk/visiondirect/ eye-gel-mask-blue Eye Gel Mask Blue placed over the closed eyes: Bag fill with temperature retention gel
  ELESTAT® (epinastine HCl ophthalmic solution) 0.05% Initial U.S. Approval: 2003 H1 histamine receptor antagonist
- No Treatment / Artificial Tear / Cold Compress: Exposure to grass pollen only
  Preservative free Hypromellose Eye Drops BP 0.3% w/v preservative free - MHRA product licence number:23097/0006 Non-Pharmaceutical Tear Supplement artificial tear
  Cooled gel eye mask http://www.visiondirect.co.uk/visiondirect/ eye-gel-mask-blue Eye Gel Mask Blue placed over the closed eyes: Bag fill with temperature retention gel
Period: Overall Study
Arm/Group | No Treatment/Artificial Tear / Cold Compress / Pharmaceutical | No Treatment / Artificial Tear / Cold Compress
Started | 11 | 7
Completed | 11 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects underwent skin prick and bilateral conjunctival challenge tests to confirm systemic and ocular allergic sensitivity to grass pollen
Groups:
- No Treatment / Artificial Tear / Cold Compress / Pharmaceutica: Exposure to grass pollen only
  Preservative free Hypromellose Eye Drops BP 0.3% w/v preservative free - MHRA product licence number:23097/0006 Non-Pharmaceutical Tear Supplement artificial tear
  Cooled gel eye mask http://www.visiondirect.co.uk/visiondirect/ eye-gel-mask-blue Eye Gel Mask Blue placed over the closed eyes: Bag fill with temperature retention gel
  ELESTAT® (epinastine HCl ophthalmic solution) 0.05% Initial U.S. Approval: 2003 H1 histamine receptor antagonist indicated for the prevention of itching associated with allergic conjunctivitis
  ELESTAT® (epinastine HCl ophthalmic solution) 0.05%: 1 drop on single occasion after exposure to grass pollen
- Total: Total of all reporting groups
Arm/Group | No Treatment / Artificial Tear / Cold Compress / Pharmaceutica | No Treatment / Artificial Tear / Cold Compress | Total
Number analyzed (Participants) | 7 | 11 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 11 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (11.0) | 29.4 (10.7) | 29.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United Kingdom | 7 | 11 | 18

OUTCOME MEASURES:

1. Primary Outcome: Symptoms
Description: Short questionnaire Ocular allergy symptomology was also measured using the eye symptom section from the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) on a 0 to 6 scale, with the summed score for itching, watering, swelling and soreness resulting in a summed score between 0 and 24. A higher score indicates a worse outcome (more severe symptoms)
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Artificial Tear Supplement: Preservative free Hypromellose Eye Drops BP 0.3% w/v preservative free - MHRA product licence number:23097/0006
  Non-Pharmaceutical Tear Supplement: artificial tear supplement (Hypromellose)
- Cold Compress: Cooled gel eye mask http://www.visiondirect.co.uk/vision-direct/eye-gel-mask-blue
  Eye Gel Mask Blue placed over the closed eyes: Bag fill with temperature retention gel
- Anti-allergic Medication: ELESTAT® (epinastine HCl ophthalmic solution) 0.05% Initial U.S. Approval: 2003 H1 histamine receptor antagonist indicated for the prevention of itching associated with allergic conjunctivitis
  ELESTAT® (epinastine HCl ophthalmic solution) 0.05%: 1 drop on single occasion after exposure to grass pollen
Arm/Group | No Treatment | Artificial Tear Supplement | Cold Compress | Anti-allergic Medication
Number analyzed (Participants) | 18 | 18 | 18 | 11
Units on a scale | 15.3 (1.8) | 11.3 (1.2) | 13.3 (1.1) | 9.8 (1.3)

2. Primary Outcome: Ocular Redness
Description: Bulbar and limbal redness will be observed with a slit lamp biomicroscope and graded using a validated scale
  • The 'Efron' grading scale consists of 5 pictures of eyes of increasing severity of blood vessels over the white of the eye, with the clinician selecting the image closest to what they observe on the patient (0 indicating a white eye and 4 a very irritated eye). There are no subscales
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Treatment | Artificial Tear Supplement | Cold Compress | Anti-allergic Medication
Number analyzed (Participants) | 18 | 18 | 18 | 11
units on a scale | 2.15 (0.40) | 1.79 (0.40) | 1.61 (0.32) | 1.78 (0.38)

3. Primary Outcome: Ocular Temperature
Description: Ocular surface temperature will be measured with an infra-red camera
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: degrees centrigrade
Arm/Group | No Treatment | Artificial Tear Supplement | Cold Compress | Anti-allergic Medication
Number analyzed (Participants) | 18 | 18 | 18 | 11
degrees centrigrade | 35.88 (0.75) | 35.91 (0.96) | 35.41 (0.88) | 34.56 (0.85)

ADVERSE EVENTS:
Arm/Group | No Treatment | Artificial Tear Supplement | Cold Compress | Anti-allergic Medication
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/11
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No